CLINICAL TRIAL: NCT00399191
Title: A Test of Iron Malabsorption in Patients With Iron Deficiency Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R43 DK64495 (completed); R43DK064495 (NIH)
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Iron Deficiency Anemia
Keywords: anemia; iron deficiency anemia; iron deficiency; absorption; iron absorption; iron uptake
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies | interventions — Dysprosium

INTERVENTIONS:
Drug: stable isotope of iron, dysprosium

SUMMARY:
The objective of the study is to develop a simple, noninvasive test for evaluation of iron absorption as a tool to determine the cause of iron deficiency anemia. Healthy, premenopausal women with iron deficiency with or without anemia will be recruited for the study. Participants will, over the course of two months, ingest an iron solution three times; after each iron ingestion, participants will collect their stool and bring it to the study investigators for assessment of iron content.

ELIGIBILITY:
Inclusion Criteria:

* ferritin <40

Exclusion Criteria:

* pregnant,
* post-partum,
* s/p GIT surgery,
* known malabsorption,
* coeliac disease,
* Helicobacter pylori

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-08

PRIMARY OUTCOMES:
initial mucosal uptake of iron
intra- and inter-individual variability
red cell incorporation of iron

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Janghorbani, PhD, Principal Investigator — BioChemAnalysis Corp.
Locations (1):
- UT Southwestern, Dallas, Texas, United States